CLINICAL TRIAL: NCT03367975
Title: NIRS Monitoring During Intracranial Interventions
Acronym: NIRS_ICG
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Bonn (Other)
Responsible Party: Principal Investigator, Martin Soehle, Consultant, University Hospital, Bonn
Other Study IDs: NIRS_039/14
Record Dates: First submitted 2014-10-03; First posted 2017-12-11 (Actual); Last update posted 2017-12-11 (Actual); Status verified 2017-12

CONDITIONS: Subarachnoid Hemorrhage; Intracranial Arteriovenous Malformation
MeSH Terms: conditions — Subarachnoid Hemorrhage; Intracranial Arteriovenous Malformations | interventions — Spectroscopy, Near-Infrared

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: near infrared spectroscopy

SUMMARY:
Near infrared spectroscopy is a valuable tool to monitor cerebral oxygenation during intracranial interventions. However, it yields artificial results when the dye indocyanine green (ICG) is applied, which is routinely done for intraoperative angiography.

The investigators examine, to what extent and which duration NIRS is disturbed following ICG application.

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled for aneurysm clipping or av-malformation removal

Exclusion Criteria:

* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing cerebral aneurysm clipping or av-malformation removal
Sampling Method: Non-Probability Sample
Enrollment: 12 (Estimated)
Dates: Start 2014-03; Primary Completion 2018-01 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
amount of rSO2 - change [%] induced by ICG-application | 1 hour
  Cerebral oxygenation (rSO2) may be quantified using NIRS. The dye ICG, that is used intraoperatively, affects NIRS, since it changes rSO2 without modifying cerebral oxygenation. The amount, by which rSO2 is altered will be assessed

CONTACTS AND LOCATIONS:
Locations (1):
- Dept. of Anaesthesiology and Intensive Care Medicine, Univ. of Bonn, Bonn, Germany